CLINICAL TRIAL: NCT04306653
Title: ACTH vs Betamethasone for the Treatment of Acute Gout in Hospitalized Patients: A Randomized, Open Label, Comparative Study
Brief Title: ACTH vs Betamethasone in Hospitalized Patients With Acute Gout
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Dimitrios Daoussis, Assoc Prof, University of Patras
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PGNP 738/17112016
Record Dates: First submitted 2020-02-14; First posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Gout Attack
Keywords: gout, ACTH
MeSH Terms: conditions — Gout | interventions — Adrenocorticotropic Hormone; Betamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACTH (Experimental): patients with acute gout treated with ACTH
  Interventions: Drug: ACTH
- Betamethasone (Active Comparator): patients with acute gout treated with betamethasone
  Interventions: Drug: Betamethasone

INTERVENTIONS:
Drug: ACTH — patients with acute gout will receive 100 IU ACTH IM
  Arms: ACTH
Drug: Betamethasone — patients with acute gout will receive 6 mg of betamethasone
  Arms: Betamethasone

SUMMARY:
Background: Hospitalized patients usually have significant comorbidities and receive multiple medications which leads to a high frequency of contraindications to standard treatment options for acute gout (NSAIDs, colchicine, steroids). Adrenocorticotropic hormone (ACTH) has long been used in acute gout, exhibiting significant clinical efficacy and an excellent safety profile. Aim: To assess 1) the clinical efficacy of ACTH in gout compared to betamethasone in hospitalized patients 2) the safety profile of ACTH vs betamethasone and 3) the effect of ACTH on immune responses and metabolic parameters. Methods: This is a randomized, open label comparative study directly comparing ACTH vs betamethasone for acute gout. The investigators plan to recruit 60 hospitalized patients who will be randomly assigned to either the ACTH or the betamethasone group on a 1:1 basis. Participants will be clinically assessed at baseline and at 24, 48, 72h and 5 days time points. (Intensity of pain, physician and patient global assessment, tenderness, swelling and redness). Serum and plasma samples will be collected at baseline and at the 24, 48, 72h time points from all study paticipants. The investigators will assess the effect of ACTH vs betamethasone on several metabolic parameters concentrating on glucose homeostasis. Results: The study is currently recruiting patients. Conclusions: If the efficacy and safety profile of ACTH is verified in this randomized controlled trial, the use of ACTH for the treatment of gout in the hospital setting will be strongly supported.

DETAILED DESCRIPTION:
BACKGROUND Treatment of gout can be either simple and straightforward in many cases, or extremely problematic in others. Current guidelines recommend the use of non-steroidal anti-inflammatory drugs (NSAIDs) and colchicine as first-line treatment. However, patients with gout typically have multiple comorbidities that often preclude the use of these drugs. The management of gout can be even more troublesome in the hospital setting. Hospitalized patients usually have significant comorbidities and receive multiple medications, which lead to a high frequency of contraindications to the above agents. Steroids are considered an alternative therapeutic option especially for "difficult-to-treat" patients such as hospitalized patients. However they associate with immunosuppression and metabolic side effects; therefore, their use in the inpatient setting may be problematic as well. Adrenocorticotropic hormone (ACTH) has long been used in gout. The interest in ACTH was revived in the mid-1990s when several studies showed that ACTH is equally effective and, in most cases, acts faster than NSAIDs and steroids and exhibits an excellent safety profile. It was previously thought that the anti-inflammatory action of ACTH was steroid related: if this was the case, then one could argue that treatment with ACTH would have no advantage over the systemic administration of steroids. However, experimental evidence challenges this view; it has been shown that ACTH mainly acts in a steroid independent manner. The investigators have been using ACTH as a first-line treatment for hospitalized patients since 1995. The investigators have reported their experience with ACTH in gout in hospitalized patients - ACTH is highly effective and associates with minimal side effects.

AIM To assess 1) the clinical efficacy of ACTH in gout compared to betamethasone in hospitalized patients; 2) the safety profile of ACTH vs betamethasone; and 3) the effect of ACTH on immune responses and metabolic parameters. HYPOTHESIS Based on retrospective data related to the use of ACTH in gout, the investigators hypothesize that ACTH has comparable clinical efficacy to betamethasone in the treatment of acute gout but exhibits a better safety profile and associates with less immunosuppression than betamethasone. STUDY DESIGN The investigators plan to recruit 60 hospitalized patients with acute gout. Participants will be randomly assigned to either the ACTH or the betamethasone group on a 1:1 basis. All participants will provide written informed consent. The study protocol has already been submitted and approved by the Ethics Committee of the University Hospital of Patras. The following data will be recorded for each participant: 1) age; 2) gender; 3) admission and discharge diagnosis; 4) history of major comorbidities that represent contraindications to established gout therapies; and 5) history history of hyperuricemia and gout. Comorbidities that will be recorded: a) hypertension defined as having a blood pressure (BP) of ≥140mmHg systolic and/or ≥90 mmHg diastolic and/or receiving any antihypertensive therapy; b) cardiovascular disease defined as the presence of coronary heart disease, cerebrovascular accident or peripheral vascular disease; c) chronic kidney disease defined as an estimated glomerular filtration rate, measured by the abbreviated Modification of Diet in Renal Disease formula of 60-90ml/min/1.73m2 (mild) or <60ml/ min/1.73m2 (moderate/severe); and d) diabetes mellitus (DM) defined as fasting serum glucose levels >126mg/ dl and/or the use of oral hypoglycemic medications or insulin. Particiopants will receive an IM injection of either 100 IU of ACTH (Synachten Depot) or 6 mg of betamethasone (Celestone Chronodose, which is the most commonly used intramuscular steroid formulation in our country and frequently used for the treatment of gout in the hospital setting. In case of partial or no response, participants will receive a second IM injection of the same drug at the 24h time point. Participants will be assessed at baseline and at 24, 48, 72h and 5-day time points. The clinical efficacy will be assessed as follows:

1. Intensity of pain will be recorded using a Visual Analogue Scale (0-10 cm) at 24, 48, 72h and 5days time points. Pain VAS will be also recorded at the 6 and 12h time points (self reported by the patient on a special diary provided);
2. Physician and patient global assessment (0-100 scale) at 24, 48, 72h and 5days time points;
3. Tenderness, swelling and redness (0-3 scale) will be recorded at 24, 48, 72h and 5days time points. LABORATORY ANALYSIS The investigators aim to assess the effects of ACTH vs betamethasone on i) metabolic parameters and ii) immune responses. i) Metabolic parameters Serum and plasma samples will be collected at baseline and at the 24, 48, 72h time points from all study participants and will be stored at -70 oC. The investigators will assess the effect of ACTH vs betamethasone on several metabolic parameters concentrating on glucose homeostasis. The invstigators propose the measurement of the following molecules in serum samples collected at the time points specified above:

1) Fasting glucose, insulin and C-peptide so we can explore the effect of ACTH vs betamethasone on glucose homeostasis; 2) Total cholesterol, LDL, HDL and triglycerides so we can explore the effect of ACTH vs betamethasone on lipid homeostasis; 3) Cortisol levels in patients treated with ACTH. So far, the effect of a single IM ACTH injection of 100IU on cortisol levels is not known. The investigators hypothesize however, that cortisol levels will raise soon following the ACTH injection and decline shortly thereafter, thus causing minimum immunosuppression. In betamethasone treated patients the investigators propose the measurement of both Cortisol (using an assay with no cross reactivity with betamethasone) and ACTH levels. The investigators hypothesize that betamethasone will have a more pronounced effect on the HPA axis than ACTH and therefore may associate with a more intense and long-lasting immunosuppression; 4) Tetracosactide (Synachten) levels and betamethasone levels in ACTH and betamethasone treated patients respectively. Tetracosactide will be measured by ELISA methodology in plasma samples (Elisa Kit from Peninsula Laboratories, San Carlos, USA) that reacts with the part 1-24 of ACTH (and thus Tetracosactide). Plasma samples will be prepared by total elimination of endogenous ACTH by cation exchange chromatography. Similarly, betamethasone levels will be measured by ELISA methodology. With these experiments the investigators will explore how long tetracosactide and betamethasone circulate in peripheral blood following a single intramuscular injection. The investigators will match these data with the data derived from the experiments presented above (cortisol levels) to explore the effect of tetracosactide (Synachten) vs betamethasone on the HPA axis. ii) Effects on immune responses The investigators will study the effects of ACTH vs betamethasone on key cells mediating immune responses, such as a) T cells and b) neutrophils. The investigators propose the study of 10 patients (5 in the ACTH and 5 in the betamethasone group) matched for age and gender. These patients will not have active infection. A) Effects on T cells The investigators will collect 20 ml of heparinized peripheral blood at baseline and at the 24h time point. Peripheral blood mononuclear cells (PBMC) will be separated using a standard Ficoll centrifugation protocol and will be immediately stored in liquid nitrogen. The investigators estimate to collect 20X106 PBMC's from each sample. When all samples have been collected, the investigators will use flow cytometry to assess the expression of several activation markers on T cells. PBMC's will be stained with fluorochrome- conjugated monoclonal antibodies against CD3, CD40L, CD69 and CD25 and their respective isotypic controls. CD40L, CD69 and CD25 are typical T cell activation markers. Flow cytometry will be used to assess the percentage of CD3+ CD40L+, CD3+ CD69+ and CD3+ CD25+ double positive cells. The investigators also propose to assess these activation markers on T cells following activation. PBMC's will be cultured in RPMI supplemented with 15% FBS and antibiotics (pen/strep) for 48h. PHA at a concentration of 1μg/ml will be added to culture medium to activate T cells. Following 48h of culture, cells will be collected by centrifugation and analyzed as above using flow cytometry. In this experiment the investigators also plan to measure IL-2 levels in the culture supernatants since IL-2 is the main cytokine produced following T cell activation. With these experiments the investigators will explore the effects of ACTH vs betamethasone on T cells which are key cells mediating adaptive immune responses. The investigators hypothesize that ACTH has less effects on T cells compared to betamethasone. If this hypothesis is conformed by the experiments presented above, it will provide indirect evidence that ACTH causes less immunosuppression than steroids. SIGNIFICANCE OF THE STUDY This will be the first study to assess the efficacy of ACTH in gout in the hospital setting in a prospective manner. The investigators have previously reported that ACTH is highly effective in these patients and exhibits an excellent safety profile; however, these data were retrospectively collected. Therefore, if the efficacy and safety profile of ACTH is verified in this randomized controlled trial, the use of ACTH for the treatment of gout in the hospital setting will be strongly supported. However, the investigators believe that the laboratory part of the study will provide even more valuable data. If ACTH is proven to cause less metabolic abnormalities and associates with less immunosuppression compared to betamethasone, then ACTH may become the treatment of choice in this setting. Considering that hospitalized patients are the most difficult-to-treat patients, this may lead to wider use of ACTH in the treatment of gout in the community as well.

ELIGIBILITY:
Inclusion Criteria:

1. Age>18 years
2. able to provide written informed consent
3. diagnosis of acute gout according to ACR/EULAR classification criteria -

Exclusion Criteria:

1. pregnancy/lactation
2. unable to provide written informed consent -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-01-05 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Pain VAS | 12 hours
  Intensity of pain will be recorded using a Visual Analogue Scale (VAS) (0-10, 0=no pain 10=worst pain)
Pain VAS | 24 hours
  Intensity of pain will be recorded using a Visual Analogue Scale (VAS) (0-10, 0=no pain 10=worst pain)
Pain VAS | 48 hours
  Intensity of pain will be recorded using a Visual Analogue Scale (VAS) (0-10, 0=no pain 10=worst pain)
Pain VAS | 72 hours
  Intensity of pain will be recorded using a Visual Analogue Scale (VAS) (0-10, 0=no pain 10=worst pain)
Pain VAS | 5 days
  Intensity of pain will be recorded using a Visual Analogue Scale (VAS) (0-10, 0=no pain 10=worst pain)

SECONDARY OUTCOMES:
Physician global assessment | 24 hours
  Physician global assessment rated on a Visual Analogue Scale (VAS) (0-100, 0=very good, 100=very bad)
Physician global assessment | 48 hours
  Physician global assessment rated on a Visual Analogue Scale (VAS) (0-100, 0=very good, 100=very bad)
Physician global assessment | 72 hours
  Physician global assessment rated on a Visual Analogue Scale (VAS) (0-100, 0=very good, 100=very bad)
Physician global assessment | 5 days
  Physician global assessment rated on a Visual Analogue Scale (VAS) (0-100, 0=very good, 100=very bad)
Patient global assessment | 24 hours
  Patient global assessment rated on a Visual Analogue Scale (VAS) (0-100, 0=very good, 100=very bad)
Patient global assessment | 48 hours
  Patient global assessment rated on a Visual Analogue Scale (VAS) (0-100, 0=very good, 100=very bad)
Patient global assessment | 72 hours
  Patient global assessment rated on a Visual Analogue Scale (VAS) (0-100, 0=very good, 100=very bad)
Patient global assessment | 5 days
  Patient global assessment rated on a Visual Analogue Scale (VAS) (0-100, 0=very good, 100=very bad)
Tenderness | 24 hours
  Tenderness rated using 0-3 scale (0=no tenderness, 3=severe tenderness)
Tenderness | 48 hours
  Tenderness rated using 0-3 scale (0=no tenderness, 3=severe tenderness)
Tenderness | 72 hours
  Tenderness rated using 0-3 scale (0=no tenderness, 3=severe tenderness)
Tenderness | 5 days
  Tenderness rated using 0-3 scale (0=no tenderness, 3=severe tenderness)
Swelling | 24 hours
  Swelling rated using 0-3 scale (0=no swelling, 3=severe swelling)
Swelling | 48 hours
  Swelling rated using 0-3 scale (0=no swelling, 3=severe swelling)
Swelling | 72 hours
  Swelling rated using 0-3 scale (0=no swelling, 3=severe swelling)
Swelling | 5 days
  Swelling rated using 0-3 scale (0=no swelling, 3=severe swelling)
Redness | 24 hours
  Redness rated using 0-3 scale (0=no redness, 3=severe redness)
Redness | 48 hours
  Redness rated using 0-3 scale (0=no redness, 3=severe redrness)
Redness | 72 hours
  Redness rated using 0-3 scale (0=no redness, 3=severe redness)
Redness | 5 days
  Redness rated using 0-3 scale (0=no redness, 3=severe redness)

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Daoussis, Principal Investigator — University of Patras Medical School
Locations (1):
- University Hospital of Patras, Pátrai, Achaia, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel LB, Alloway JA, Nashel DJ. Comparison of adrenocorticotropic hormone and triamcinolone acetonide in the treatment of acute gouty arthritis. J Rheumatol. 1994 Jul;21(7):1325-7. PMID 7966077
- [Background] Axelrod D, Preston S. Comparison of parenteral adrenocorticotropic hormone with oral indomethacin in the treatment of acute gout. Arthritis Rheum. 1988 Jun;31(6):803-5. doi: 10.1002/art.1780310618. PMID 2454635
- [Background] Ritter J, Kerr LD, Valeriano-Marcet J, Spiera H. ACTH revisited: effective treatment for acute crystal induced synovitis in patients with multiple medical problems. J Rheumatol. 1994 Apr;21(4):696-9. PMID 8035395
- [Background] Getting SJ, Christian HC, Flower RJ, Perretti M. Activation of melanocortin type 3 receptor as a molecular mechanism for adrenocorticotropic hormone efficacy in gouty arthritis. Arthritis Rheum. 2002 Oct;46(10):2765-75. doi: 10.1002/art.10526. PMID 12384937
- [Background] Getting SJ, Lam CW, Chen AS, Grieco P, Perretti M. Melanocortin 3 receptors control crystal-induced inflammation. FASEB J. 2006 Nov;20(13):2234-41. doi: 10.1096/fj.06-6339com. PMID 17077300
- [Background] Daoussis D, Antonopoulos I, Yiannopoulos G, Andonopoulos AP. ACTH as first line treatment for acute gout in 181 hospitalized patients. Joint Bone Spine. 2013 May;80(3):291-4. doi: 10.1016/j.jbspin.2012.09.009. Epub 2012 Nov 26. PMID 23195793
- [Background] Mitroulis I, Kambas K, Chrysanthopoulou A, Skendros P, Apostolidou E, Kourtzelis I, Drosos GI, Boumpas DT, Ritis K. Neutrophil extracellular trap formation is associated with IL-1beta and autophagy-related signaling in gout. PLoS One. 2011;6(12):e29318. doi: 10.1371/journal.pone.0029318. Epub 2011 Dec 16. PMID 22195044
- [Background] Gavillet M, Martinod K, Renella R, Harris C, Shapiro NI, Wagner DD, Williams DA. Flow cytometric assay for direct quantification of neutrophil extracellular traps in blood samples. Am J Hematol. 2015 Dec;90(12):1155-8. doi: 10.1002/ajh.24185. Epub 2015 Oct 6. PMID 26347989
- [Result] Khanna D, Fitzgerald JD, Khanna PP, Bae S, Singh MK, Neogi T, Pillinger MH, Merill J, Lee S, Prakash S, Kaldas M, Gogia M, Perez-Ruiz F, Taylor W, Liote F, Choi H, Singh JA, Dalbeth N, Kaplan S, Niyyar V, Jones D, Yarows SA, Roessler B, Kerr G, King C, Levy G, Furst DE, Edwards NL, Mandell B, Schumacher HR, Robbins M, Wenger N, Terkeltaub R; American College of Rheumatology. 2012 American College of Rheumatology guidelines for management of gout. Part 1: systematic nonpharmacologic and pharmacologic therapeutic approaches to hyperuricemia. Arthritis Care Res (Hoboken). 2012 Oct;64(10):1431-46. doi: 10.1002/acr.21772. No abstract available. PMID 23024028
- [Result] Keenan RT, O'Brien WR, Lee KH, Crittenden DB, Fisher MC, Goldfarb DS, Krasnokutsky S, Oh C, Pillinger MH. Prevalence of contraindications and prescription of pharmacologic therapies for gout. Am J Med. 2011 Feb;124(2):155-63. doi: 10.1016/j.amjmed.2010.09.012. PMID 21295195
- [Result] Daoussis D, Antonopoulos I, Andonopoulos AP. ACTH as a treatment for acute crystal-induced arthritis: update on clinical evidence and mechanisms of action. Semin Arthritis Rheum. 2014 Apr;43(5):648-53. doi: 10.1016/j.semarthrit.2013.09.006. Epub 2013 Oct 5. PMID 24762710
- [Derived] Daoussis D, Kordas P, Varelas G, Michalaki M, Onoufriou A, Mamali I, Iliopoulos G, Melissaropoulos K, Ntelis K, Velissaris D, Tzimas G, Georgiou P, Vamvakopoulou S, Paliogianni F, Andonopoulos AP, Georgopoulos N. ACTH vs steroids for the treatment of acute gout in hospitalized patients: a randomized, open label, comparative study. Rheumatol Int. 2022 Jun;42(6):949-958. doi: 10.1007/s00296-022-05128-x. Epub 2022 Apr 21. PMID 35445840